CLINICAL TRIAL: NCT04283734
Title: Usefulness of the Use of Co-registration Strategy With iFR in Long and/or Diffuse Coronary Lesions
Acronym: iLARDI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iLARDI
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Instantaneous Wave Free Ratio; Diffuse Coronary Artery Disease; Long Coronary Lesion; Syncvision Software
Keywords: Diffuse coronary artery disease; Instantaneous Wave Free Ratio; Long coronary lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Long/diffuse coronary lesion should be evaluated and guided by iFR pullback with Syncvision software to achieve a final iFR of 0.90
  Interventions: Device: iFR pullback with Syncvision software (Volcano company)
- Control group (No Intervention): Long/diffuse coronary lesion should be treated guided by angiography

INTERVENTIONS:
Device: iFR pullback with Syncvision software (Volcano company) — iFR pullback with Syncvision software permit us to analyze the vessel completely and to predict the physiological significance of every lesion and segment, to predict the benefit of the revascularization in terms of iFR improvement, and to predict the minimum stent length necessary to achieve this improvement.
  Arms: Intervention group

SUMMARY:
Randomized controlled trial to determinate if the physiological iFR pullback evaluation with Syncvision software (intervention group) could be useful in the reduction of stent length implanted, with the potencial benefit in terms of MACEs reduction at follow-up with respect to angiographic guiding of percutaneous coronary intervention (control group).

DETAILED DESCRIPTION:
Physiological coronary lesion evaluation is actually a routine practice in the labs to guide percutaneous coronary intervention decision making. Unlike FFR, the new index permit us to perform an analysis of the physiological importance of every lesion and every coronary segment. This fact has allowed to create a new specific software. Syncvision show us the functional compromise of every lesion and predict the expected IFR improvement.

This potential benefit could have an extra benefit in the reduction of the implanted stent length. There are some observational study published that reported a reduction of 5 mm of stent length, but we think that the reduction could be significantly higher.

However, this reduction could be detrimental of the complete cover of plaque in this type of lesion, which has also proved to be a predictor of MACEs.

For this reason, we have proposed to perform a randomized study to define if the utilization of physiological IFR pullback evaluation in long and/or diffuse coronary lesion present advantages over classical angiographic PCI.

Study hyphotesis:

Revascularization guided by IFR-Pullback in long and/or diffuse coronary lesions permit to reduce the stent length implanted, with the potential benefit in terms of MACEs reduction.

Study design:

Randomized and controlled study where we will include patients with significant coronary stenosis at least in one vessel and a total lesion length higher than 30 mm in the different clinical scenarios (stable angina, NSTEMI and STEMI in non-culprit lesion).

In the control group, stent length will be decided by the operator. In the iFR-pullback group, stent length will be decided in base to iFR expected, trying to obtain an IFR of 0.90 with the minimum stent length as possible.

The expected stent length reduction is 15 mm (primary endpoint). As secondary endpoint, we will analyze the combined endpoint of myocardial infarction, death and new revascularization).

The sample size in base to primary endpoint will be of 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age higher than 18 years old.
* Sign of inform consent
* Patients with at least a vessel with angiographic significant lesion (long/sequential or diffuse lesion) >/= 25 mm of length where the percutaneous strategy is going to be the choice strategy.
* Patients with stable angina, NSTEMI or STEMI (non culprit vessel)

Exclusion Criteria:

* Patients with Acute Coronary Syndrome with non optimal result of culprit vessel (final TIMI flow < TIMI III, non-reflow phenomenon during the treatment, residual coronary dissection, lost or compromise of significant side branch).
* Acute Coronary Syndrome and Left Ventricular Ejection Fraction lower than 45%.
* Live expectancy lower than 12 months.
* Patients with severe aortic stenosis.
* Contraindication for dual anti platelet therapy during at least 12 months.
* Patients with indication of bypass surgery in base to Heart Team decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2024-01-24 (Estimated); Study Completion 2024-01-24 (Estimated)

PRIMARY OUTCOMES:
Reduction of the average stent length implanted in the Syncvision guided group | 12 months
  Reduction of stent length implanted, measured in millimeters, in the group guided by Syncvision software

SECONDARY OUTCOMES:
Combined endpoint of cardiac death, myocardial infarction and new revascularization of analyzed or treated vessel in the basal procedure at 12 months of follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Hidalgo, PhD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The shared documents will be available after the publication for 1 year.
Access Criteria: By e-mail to uicec@imibic.org

REFERENCES:
- [Derived] Hidalgo F, Gonzalez-Manzanares R, Suarez de Lezo J, Gallo I, Alvarado M, Perea J, Maestre-Luque LC, Resua A, Romero M, Lopez-Benito M, Perez de Prado A, Ojeda S, Pan M. The Usefulness of Coregistration with iFR in Tandem or Long Diffuse Coronary Lesions: The iLARDI Randomized Clinical Trial. J Clin Med. 2024 Jul 25;13(15):4342. doi: 10.3390/jcm13154342. PMID 39124613